CLINICAL TRIAL: NCT02734641
Title: Does Increase in Appetite After Iron Treatment Induced by Ghrelin Hormone
Status: Completed | Type: Observational
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Sponsor
Other Study IDs: 155-15EMC
Record Dates: First submitted 2016-02-04; First posted 2016-04-12 (Estimated); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- intravenous (IV) iron therapy: Patients register to intravenous (IV) iron therapy due to iron deficiency anemia that wasn't responded to oral treatment or wasn't tolerable due to side effects.
  20 mL of blood will be draw for complete blood count, renal function, electrolytes and ghrelin. In addition, the patient will fill a structured questionnaire that examines the appetite of the patient before and after treatment. At the end of Iron administration Ghrelin will be retested.
- healthy volunteer: healthy volunteer, will be asked 20 mL of blood will be draw for complete blood count, renal function, electrolytes and ghrelin. In addition, the patient will fill a structured questionnaire that examines his appetite. Ghrelin will be retested after 6 weeks.

SUMMARY:
The purpose of this study is to examine whether iron therapy in patients with intravenous iron deficiency anemia causes an increase in appetite. And whether this increase is mediated by the hormone ghrelin.

DETAILED DESCRIPTION:
Prior to Iron treatment Investigator will sample subject blood for: counting blood, iron sector indices, renal function, electrolytes, and measure the level of ghrelin fasting plasma. In addition, the patient will fill a structured questionnaire that examines appetite levels. participants will be asked to answer a structured questionnaire which will include information on demographics, clinical data (fever, allergies, weight, height) and comorbidities. Additional data on laboratory tests, comorbidities, medication and regular blood and urine cultures results will be taken from the medical file. Iron treatment will be given according to local standard procedure . At the end of the treatment ghrelin levels and questionaire will be retaken .

iron deficiency anemia is defined: hemoglobin <12 gr / dl in women and Hb <13 gr / dl in men with ferritin <15 ng / ml.

ELIGIBILITY:
Inclusion Criteria:

* Iron deficiency anemia that wasn't responded to oral treatment or wasn't tolerable due to side effects
* sign and dated informed consent form.

Exclusion Criteria:

* chronic inflammatory disease.
* chronic renal failure
* active cancer.
* active Infectious disease.
* non iron deficiency anemia.
* pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients register to intravenous (IV) iron therapy due to iron deficiency anemia that wasn't responded to oral treatment or wasn't tolerable due to side effects and healthy volunteer.
Sampling Method: Probability Sample
Enrollment: 111 (Actual)
Dates: Start 2016-08; Primary Completion 2017-04-01 (Actual); Study Completion 2018-04-17 (Actual)

PRIMARY OUTCOMES:
Ghrelin levels after treatment with Intravenous Iron | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: mazen Elias, prof, Principal Investigator — HaEmek Medical Center, Israel
Locations (1):
- Haemek medical center, Afula, Israel

IPD SHARING:
Plan to Share IPD: Undecided